CLINICAL TRIAL: NCT04076813
Title: Cangrelor in Acute Myocardial Infarction: Effectiveness and Outcomes Registry
Acronym: CAMEO
Status: Active, not recruiting | Type: Observational
Sponsor: Chiesi USA, Inc. (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00100421
Record Dates: First submitted 2019-08-30; First posted 2019-09-03 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Myocardial Infarction
Keywords: cangrelor
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- STEMI/NSTEMI: Patients in the registry will be 18 years of age or older and underwent coronary angiography for a ST-elevation myocardial infarction (STEMI) or NSTEMI Non-ST-elevation myocardial infarction

SUMMARY:
The purpose of this registry is to address optimal platelet inhibition during the early management of MI patients prior to coronary angiography or CABG.

DETAILED DESCRIPTION:
The CAMEO registry is a multicenter observational registry that will collect information on approximately 5,050 patients with NSTEMI or STEMI treated with cangrelor or an oral P2Y12 inhibitor into the registry.

Phase 1: Each site will abstract data from the medical record for the first 50 patients meeting the inclusion and exclusion criteria treated at the hospital within 4 months prior to study initiation or during the study period.

Phase 2: After Phase 1, all cangrelor-treated patients meeting the inclusion and exclusion criteria will be entered into the registry, and we will begin sampling non-cangrelor patients in a 2:1 cangrelor: non-cangrelor ratio (Phase 2) up to 3000 patients.

Phase 3: We will work with sites on a quality improvement initiative with the current sites to 1) continue enrollment of an additional 2,000 patients; 2) provide feedback reports to both the sites and operators about the use and administration of cangrelor to patients they are treating; 3) utilize a pharmacist-based group with representatives from each site to identify opportunities to improve use of cangrelor according to the established treatment strategy.

ELIGIBILITY:
Phase 1 Inclusion Criteria:

For the first 50 patients at each participating site, consecutive patients are entered in the registry if they are ≥ 18 years of age, underwent coronary angiography for a STEMI or NSTEMI, and received cangrelor at any time during the hospitalization or an oral P2Y12 inhibitor during his/her first 48 hours of the hospitalization for MI.

Phase 2 Inclusion Criteria:

Subsequent patients are eligible to be entered in the registry if they are ≥ 18 years of age and underwent coronary angiography for a STEMI or NSTEMI and meet at least 1 of the following criteria:

1. The patient was hospitalized for STEMI and met one of the following inclusion criteria:

   * The patient received cangrelor at any time during his/her hospitalization for MI.
   * The patient received an oral P2Y12 inhibitor during his/her first 48 hours of hospitalization AND either of the following:
   * The patient received a P2Y12 inhibitor and an opiate/opioid within 24 hours prior to or during primary PCI for STEMI presentation.

   OR
   * The patient underwent coronary angiography followed by CABG during the index MI admission and received any P2Y12 inhibitor within 7 days prior to CABG.
2. The patient was hospitalized for NSTEMI and met one of the following inclusion criteria:

   * The patient received cangrelor during his/her hospitalization for MI.
   * The patient received an oral P2Y12 inhibitor during his/her first 48 hours of hospitalization AND either of the following:
   * The patient underwent coronary angiography followed by CABG during the index MI admission and received any P2Y12 inhibitor within 7 days prior to CABG. OR
   * Any 2 of the following criteria without prior PCI or CABG: age> 60 years, male sex, diabetes, EF <40% prior heart failure

Exclusion Criteria: If the patient does not meet the inclusion criteria for either Phase.

Phase 3 Eligibility Criteria:

The Phase 3 portion of the CAMEO registry will focus on launching local site quality improvement initiatives with the goal of optimizing cangrelor usage according to FDA-approved established treatment strategy. Enrollment for the registry will be extended for an additional two years to include an additional 2,000 patients in this phase of the registry. The inclusion criteria of these patients will be the same as in Phase 2 (see section 3.3.2). We will also capture which patients are cared for at each site by individual operators. Operator-level data will be de-identified, and each operator will be assigned an operator ID. Sites will be asked to maintain a crosswalk for operator ID, and complete an operator characteristics survey. The operator characteristics survey will ask questions around age, sex, and other relevant operator characteristics, and will be used in the analysis phase in aggregate. Operators will not be directly identified and the analytics center will not have access to the crosswalk, which will be maintained at the site.

We will identify a pharmacist representative at each site to form a pharmacist-based group who meets monthly to identify strategies to improve processes at each site and to improve use of cangrelor in the MI population according to the established treatment strategy. We will present quarterly feedback reports to the sites that include data regarding the use of cangrelor according to the following parameters: 1) administration of both a bolus and infusion; 2) appropriate timing between infusion and initiation of oral PY212 inhibitor therapy; 3) and administration of the infusion based on clinical trial data and dose package labeling for patients who are able to be transitioned to oral P2Y12 inhibitor therapy shortly after PCI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ≥ 18 years of age and underwent coronary angiography for a STEMI or NSTEMI.
Sampling Method: Probability Sample
Enrollment: 5050 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The number of Antiplatelet medications used during hospitalization | The time frame is hospitalization through discharge, approximately 3 days
  Antiplatelet use, including switching and discontinuation will be measured by medical record report. The medical record report will include medication start and stop dates and times.
Number of bleeding events during hospitalization as measured by medical record report | The time frame is hospitalization, up to 7 days post discharge
  Bleeding event entered from the medical record report.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rymer, MD, Principal Investigator — Duke University; Jeffrey Washam, Principal Investigator — Duke University
Locations (11):
- United States (11):
  - The Regents of the University of California on behalf of its San Diego campus, La Jolla, California
  - Christiana Care Health Services, Inc., Newark, Delaware
  - University of Florida, Gainesville, Florida
  - Kootenai Hospital District dba Kootenai Health, Coeur d'Alene, Idaho
  - MedStar Health Research Institute, Inc., Hyattsville, Maryland
  - The Brigham and Women's Hospital, Inc., Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - The Trustees of Columbia University in the City of New York, New York, New York
  - Duke University, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
There is not a current plan to share IPD.

REFERENCES:
- [Background] Rymer JA, Bhatt DL, Angiolillo DJ, Diaz M, Garratt KN, Waksman R, Edwards L, Tasissa G, Salahuddin K, El-Sabae H, Dell'Anna C, Davidson-Ray L, Washam JB, Ohman EM, Wang TY. Cangrelor Use Patterns and Transition to Oral P2Y12 Inhibitors Among Patients With Myocardial Infarction: Initial Results From the CAMEO Registry. J Am Heart Assoc. 2022 Jun 7;11(11):e024513. doi: 10.1161/JAHA.121.024513. Epub 2022 May 27. PMID 35621210
- [Background] Rymer J, Alhanti B, Kemp S, Bhatt DL, Kochar A, Angiolillo DJ, Diaz M, Garratt KN, Wimmer NJ, Waksman R, Kirtane AJ, Ang L, Bach R, Barker C, Jenkins R, Basir MB, Sullivan A, El-Sabae H, Brothers L, Ohman EM, Jones WS, Washam JB, Wang TY. Risk of Bleeding Among Cangrelor-Treated Patients Administered Upstream P2Y12 Inhibitor Therapy: The CAMEO Registry. J Soc Cardiovasc Angiogr Interv. 2023 Nov 27;3(2):101202. doi: 10.1016/j.jscai.2023.101202. eCollection 2024 Feb. PMID 39132213
- [Background] Rymer J, Pichan C, Page C, Alhanti B, Bhatt DL, Kochar A, Angiolillo DJ, Diaz M, Wimmer NJ, Waksman R, Ang L, Bach R, Jenkins R, El-Sabae H, Brothers L, Ohman EM, Jones WS, Washam JB, Wang TY, Narcisse D, Basir MB. The Use of Cangrelor in Cardiogenic Shock: Insights from the CAMEO Registry. J Card Fail. 2024 Oct;30(10):1233-1240. doi: 10.1016/j.cardfail.2024.08.003. PMID 39389732